CLINICAL TRIAL: NCT07307703
Title: Effects of Transcutaneous Electrical Nerve Stimulation (TENS) on Surgical Anxiety, Postoperative Pain, and Patient Satisfaction in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: TENS for Anxiety, Pain, and Satisfaction After Laparoscopic Cholecystectomy
Acronym: TENS-LC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Abdurrahman Acar, Research Assistant, Faculty of Health Sciences, Niğde Ömer Halisdemir University, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22504254-050.04Cholecystectomy
Record Dates: First submitted 2025-12-10; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Gallstone Disease; Postoperative Pain; Surgical Anxiety; Patient Satisfaction After Laparoscopic Cholecystectomy
Keywords: Laparoscopic Cholecystectomy; Gallstone Disease; Surgical Anxiety; Postoperative Pain; Transcutaneous Electrical Nerve Stimulation (TENS)
MeSH Terms: conditions — Cholelithiasis; Pain, Postoperative | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model. Participants undergoing elective laparoscopic cholecystectomy will be randomly assigned to one of two groups:
  Intervention group: Patients will receive Transcutaneous Electrical Nerve Stimulation (TENS) in addition to standard perioperative care.
  Control group: Patients will receive standard perioperative care without TENS.
Masking Description: No additional parties are masked in this study. Due to the nature of the intervention (TENS), participants and care providers are aware of group allocation. The study is conducted as an open-label randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 TENS Group (Experimental): Participants in this arm will receive Transcutaneous Electrical Nerve Stimulation (TENS) in addition to standard perioperative care for laparoscopic cholecystectomy. TENS will be applied using surface electrodes placed on intact skin before and after surgery. The stimulation parameters will follow established clinical guidelines to ensure safety and effectiveness. Outcomes assessed include surgical anxiety, postoperative pain intensity, and patient satisfaction.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Control Group (No Intervention): Participants in this arm will receive standard perioperative care for laparoscopic cholecystectomy without Transcutaneous Electrical Nerve Stimulation (TENS). Usual surgical and nursing protocols will be followed according to hospital standards. Outcomes assessed include surgical anxiety, postoperative pain intensity, and patient satisfaction, which will be compared with the intervention group to evaluate the added effect of TENS.

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Transcutaneous Electrical Nerve Stimulation (TENS) is a non-invasive device-based intervention that delivers mild electrical currents through electrodes placed on intact skin. In this study, TENS will be applied perioperatively to patients undergoing laparoscopic cholecystectomy. The stimulation sessions will be conducted before and after surgery, following standardized clinical parameters to ensure safety and reproducibility. The intervention is designed to evaluate its effects on surgical anxiety, postoperative pain intensity, and patient satisfaction compared with standard care.
  Other Names: TENS Therapy; Electrical Nerve Stimulation
  Arms: Arm 1 TENS Group

SUMMARY:
This study is designed to evaluate whether Transcutaneous Electrical Nerve Stimulation (TENS) can improve recovery for patients undergoing laparoscopic gallbladder removal surgery (laparoscopic cholecystectomy). TENS is a non-invasive method that uses mild electrical currents applied through the skin to stimulate nerves.

The main goals of the study are to determine if TENS can:

Reduce surgical anxiety before and during the procedure

Decrease postoperative pain after surgery

Improve overall patient satisfaction with their surgical experience

Patients who participate will receive standard surgical care, and some will also receive TENS therapy. Outcomes will be measured using patient questionnaires and clinical assessments during the hospital stay and follow-up period.

By comparing patients who receive TENS with those who do not, the study aims to provide evidence on whether this simple technique can enhance comfort and recovery after gallbladder surgery.

DETAILED DESCRIPTION:
Gallstone disease is common in Western countries, and cholecystectomy is a routine abdominal surgical procedure. The laparoscopic approach is considered the gold standard. However, many patients experience acute postoperative pain, often reported as moderate to severe. Acute pain delays recovery and may lead to complications.

Opioids remain the cornerstone of postoperative pain management, but they are associated with adverse effects such as sedation, nausea, respiratory depression, and opioid-induced hyperalgesia. In addition, long-term problematic opioid use has been reported in 6-8% of patients after surgery. Therefore, non-pharmacological alternatives for postoperative pain relief are urgently needed.

Transcutaneous Electrical Nerve Stimulation (TENS) is a non-invasive intervention that delivers electrical currents through electrodes placed on intact skin. Evidence from systematic reviews and meta-analyses suggests that TENS is effective and safe for managing both acute and chronic pain, with minimal side effects and low cost. Patients may experience mild tingling or discomfort, and rarely skin irritation.

Despite promising data, few studies have evaluated the combined effects of TENS on surgical anxiety, postoperative pain, and patient satisfaction in laparoscopic cholecystectomy. Most prior research has focused only on pain outcomes, neglecting psychological dimensions and patient-centered measures. This study aims to fill that gap by assessing whether TENS can reduce perioperative anxiety, improve pain control, and enhance satisfaction with surgical care.

This randomized controlled trial will be conducted at Adana City Training and Research Hospital between October 2025 and October 2026. Eligible patients undergoing elective laparoscopic cholecystectomy will be randomized into two groups: a TENS intervention group and a control group receiving standard care. The sample size was determined by power analysis, requiring 40 participants per group (total n=80).

Data collection will include:

Personal Information Form (demographics and baseline characteristics)

Visual Analog Scale (VAS) for pain intensity

Surgery-Specific Anxiety Scale (validated Turkish instrument)

Newcastle Satisfaction with Nursing Care Scale (validated Turkish version)

Exclusion criteria include emergency cholecystectomy, conversion to open surgery, presence of pacemakers or implanted devices, uncontrolled epilepsy, chronic opioid use, severe psychiatric or cognitive disorders, dermatological contraindications, or concurrent participation in another clinical trial.

The primary outcomes are surgical anxiety, postoperative pain, and patient satisfaction. Secondary outcomes include recovery parameters and adverse events.

Hypotheses:

Null hypothesis (H0): TENS has no effect on surgical anxiety, postoperative pain, or patient satisfaction in laparoscopic cholecystectomy.

Alternative hypothesis (H1): TENS reduces surgical anxiety and postoperative pain while increasing patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years scheduled for elective laparoscopic cholecystectomy

ASA (American Society of Anesthesiologists) physical status classification I-II

Ability to understand the study procedures and provide written informed consent

No contraindications to TENS application (e.g., intact skin at electrode placement sites)

Willingness to comply with perioperative assessments (pain, anxiety, satisfaction scales)

Exclusion Criteria:

* Patients with ASA III or higher physical status

Presence of cardiac pacemaker or other implanted electrical devices

History of epilepsy, severe neuropathy, or psychiatric disorders affecting pain/anxiety perception

Skin lesions, infections, or dermatological conditions at electrode placement sites

Use of analgesics, anxiolytics, or sedatives beyond standard perioperative protocols

Emergency cholecystectomy or conversion to open surgery

Pregnant or breastfeeding women

Patients unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity (VAS) | Within the first 24 hours after surgery
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a validated 10 cm scale ranging from 0 (no pain) to 10 (worst imaginable pain). Patients will be asked to mark their pain level at specified postoperative intervals. The primary analysis will compare mean pain scores between the TENS group and the control group to determine whether TENS reduces postoperative pain following laparoscopic cholecystectomy.
Postoperative Pain Intensity | Within the first 24 hours after surgery
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a validated 10 cm scale ranging from 0 (no pain) to 10 (worst imaginable pain). Patients will be asked to mark their pain level at specified postoperative intervals. The primary analysis will compare mean pain scores between the TENS group and the control group to determine whether TENS reduces postoperative pain following laparoscopic cholecystectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Adana City Hospital, Niğde, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves a limited sample size and is conducted at a single institution. Ethical considerations and institutional policies restrict the sharing of raw patient-level data. Only aggregated results will be reported in publications.